CLINICAL TRIAL: NCT05595954
Title: Impact of Personalised Cardiac Anaesthesia and Cerebral Autoregulation on Neurological Outcomes in Patients Undergoing Cardiac Surgery (PRECISION)
Brief Title: Impact of Personalised Cardiac Anaesthesia and Cerebral Autoregulation on Neurological Outcomes in Patients Undergoing Cardiac Surgery
Acronym: PRECISION
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-01457; am22Gomes
Record Dates: First submitted 2022-10-18; First posted 2022-10-27 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Delirium; Postoperative Stroke; Postoperative Cognitive Dysfunction
Keywords: cerebral autoregulation; hypotension; neurological outcomes; adverse neurological events; postoperative delirium; postoperative stroke; postoperative cognitive decline; personalised cardiac anaesthesia; cardiac surgery; near-infrared spectroscopy; transcranial Doppler
MeSH Terms: conditions — Emergence Delirium; Postoperative Cognitive Complications; Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The remaining biological materials (non-genetic and genetic) will be stored in biobanks in accordance with local technical and legal standards for 10 years after publication of this study for future research projects that have not yet been defined in more detail and for which a ethical approval will be attained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Preoperative data collection — Preoperatively, patients will be assessed with Montreal Cognitive Assessment (MoCA), Geriatric Depression Scale (GDS), Clinical Frailty Scale, 3-minute Diagnostic interview for Confusion Assessment Method-defined delirium (3D-CAM, incl. severity score), modified National Institutes of Health Stroke Scale (mNIHSS), and hand grip strength measurement (using a hand dynamometer) to establish a baseline measurement of the physical, cognitive and mental status.
Diagnostic Test: Intraoperative NIRS — Intraoperatively, NIRS data will be collected and recorded in real-time.
Diagnostic Test: Intraoperative TCD — Intraoperatively, TCD data will be collected and recorded in real-time.
Diagnostic Test: Intraoperative invasive MAP — Intraoperatively, invasive arterial blood pressure data will be collected and recorded in real-time.
Diagnostic Test: Postoperative NIRS — Postoperatively, NIRS monitoring will be continued in the ICU after the surgery until (i) endotracheal extubation, or (ii) for the first 24 hours or (iii) until emergency re-operation, whichever occurs first.
Other: Postoperative data collection — Postoperatively patients will be evaluated for POD with 3D-CAM or CAM-ICU and for clinical stroke with mNIHSS. Postoperative neurocognitive disorders will be assessed using MoCA.
Diagnostic Test: Collection of serum biomarker panel — The serum biomarker panel will consist, at least, of four markers of neurological injury glial fibrillary acidic protein (GFAP), neurofilament light chain (NfL), total tau and ubiquitin-carboxy-terminal hydrolase-L1 (UCH-L1). Blood samples will be obtained preoperatively, after ICU admission, on postoperative day 1, 2, 6 (or hospital discharge, whichever occurs first) and between 6 and 12 weeks after surgery.
Diagnostic Test: Collection of blood sample for genetic study — A blood sample for the genetic study will be obtained preoperatively.

SUMMARY:
This international, multicentre prospective cohort study will assess whether perioperative duration and magnitude of mean arterial pressure (MAP) outside of an individual's cerebral autoregulation (CA) limits using near-infrared spectroscopy (NIRS) and transcranial Doppler (TCD) are associated with adverse neurological events. It is to investigate whether patients with a higher burden of cerebral haemodynamic insults have an increased incidence or poorer neurological outcomes. Associations between neurologic outcomes, neurobiomarkers and genetic tests will be explored.

DETAILED DESCRIPTION:
Adverse neurological events include perioperative neurocognitive disorders and stroke and remain one of the major risks after cardiac surgery. A lack of a comprehensive knowledge of their causes and neuroprotective strategies has hindered the development of strategies to effectively reduce these complications. Against this background, this research project will take three approaches. First, non-invasive, personalised cerebral autoregulation-oriented blood pressure monitoring aims to reduce complications by uncovering blood pressure targets tailored to individual characteristics. In parallel, establishing biological associations between adverse neurological outcomes, brain injury biomarkers and genetic studies are complementary strategies that make a move to a proactive patient-tailored paradigm, ultimately understanding the mechanisms and improving patient outcomes, patient safety and quality of life.

Therefore, this international, multicentre prospective cohort study will assess whether perioperative duration and magnitude of MAP outside of an individual's CA limits using NIRS and TCD are associated with adverse neurological events. It is to investigate whether patients with a higher burden of cerebral haemodynamic insults, defined by the duration and magnitude spent outside of an individual's CA limits based on NIRS and/or TCD, have an increased incidence of postoperative delirium (POD), stroke or cognitive decline. Biological associations between adverse neurological outcomes, the role of brain injury serum biomarkers will be explored. Genetic studies will be conducted on participants who give written informed consent for these further investigations.

ELIGIBILITY:
Inclusion Criteria:

* Elective primary or reoperative coronary artery bypass graft and/or valvular and/or ascending aorta surgery requiring cardiopulmonary bypass.

Exclusion Criteria:

* Surgery requiring moderate (28-31.9ºC) or deep (<28ºC) hypothermic circulatory arrest;
* Heart and/or lung transplantation;
* Urgent (within 24 hours) and emergency surgery;
* Inability to follow procedures or insufficient knowledge in English, German or French;
* Inability to give consent.

Participants who undergo cardiac surgery under minimal extracorporeal circulation will also be excluded.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The target population consists of in-hospital patients undergoing cardiac surgery at three centres in two European countries. Patients will be screened for eligibility. Therefore, consecutive ongoing recruitment of patients fulfilling the in- and exclusion criteria will take place during daily clinical practice at the participating hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change in 3D-CAM to assess postoperative delirium (POD) | Assessed daily on postoperative days 0 to 7 (or up to discharge, whichever occurs earlier)
  Change in 3D-CAM to assess POD. The 3D-CAM rates four diagnostic features, including acute onset and fluctuating course, inattention, disorganized thinking, and altered level of consciousness. Delirium scored as 'present' (1) or 'absent' (0) based on question responses.
Change in Confusion Assessment Method for the ICU (CAM-ICU) to assess postoperative delirium (POD) | Assessed daily on postoperative days 0 to 7 (or up to discharge, whichever occurs earlier)
  CAM-ICU is an adaptation of the CAM to be usable by clinicians to screen for delirium in the intensive care unit setting designed for intubated patients. The CAM-ICU utilizes the CAM diagnostic algorithm. There are four core features including acute onset or fluctuating course, inattention, disorganized thinking, and altered level of consciousness rated with 8 items. 3 of the 4 features must be present for CAM-ICU to be considered positive, according to the original CAM algorithm. Items are rated absent/present base on specific thresholds.

SECONDARY OUTCOMES:
Change in modified National Institutes of Health Stroke Scale (mNIHSS) | Assessed daily on postoperative days 0 to 7 (or up to discharge, whichever occurs earlier)
  Change in mNIHSS to assess postoperative clinical stroke
Change in Montreal Cognitive Assessment (MoCA) | Between 6 weeks and 12 weeks, and up to 12 months after surgery
  Change in MoCA to assess postoperative neurocognitive disorder
Postoperative increase in serum creatinine | Within 48 hours after surgery
  Postoperative increase in serum creatinine of ≥ 26.5 μmol/l (≥ 0.3 mg/dl) within 48 hours or ≥ 1.5 times of baseline to assess acute kidney injury
De novo renal replacement therapy | Within postoperative day 7 (or up to discharge)
  De novo renal replacement therapy
Major morbidity | Within postoperative day 7 (or up to discharge)
  Major morbidity as defined by the Society of Thoracic Surgeons as having at least one of the following adverse outcomes: stroke, surgical re-exploration for any cardiac reason (bleeding, coronary graft occlusion, valve dysfunction, and others), renal failure, deep sternal wound infection/mediastinitis, and prolonged ventilation (> 24 hours)
Intensive care unit (ICU) stay (in hours) | From day of surgery until discharge from ICU (approx. 1 day)
  Number of hours in ICU
Length of hospital stay (in days) | From day of surgery until discharge from hospital (approx. 7 days)
  Number of days in hospital
Perioperative mortality | Within within 30 days after surgery
  Perioperative mortality, defined as any in-hospital or postdischarge death within 30 days after surgery, regardless of cause, or any death occurring during the hospitalisation, even after 30 days
Change in brain injury biomarker panel | At preoperative screening; at day of surgery; at postoperative day 1, 2 and 6 (or hospital discharge, whichever occurs first); between 6 weeks and 12 weeks after surgery
  The serum biomarker panel consists of at least four markers of neurological injury: glial fibrillary acidic protein (GFAP), neurofilament light (NfL), total tau, and ubiquitin-carboxy-terminal hydrolase-L1 (UCH-L1).

CONTACTS AND LOCATIONS:
Overall Officials: Nuno V. Gomes, MD, Principal Investigator — Clinic for Anaesthesia, Intermediate Care, Prehospital Emergency Medicine and Pain Therapy, University Hospital Basel
Locations (4):
- Switzerland (2):
  - Clinic for Anaesthesia, Intermediate Care, Prehospital Emergency Medicine and Pain Therapy, University Hospital Basel, Basel
  - Inselspital, Bern University Hospital, Bern
- United Kingdom (2):
  - Cambridge University Hospitals and Brain Physics Lab, Cambridge
  - Royal Papworth Hospital, Department of Anaesthesia and Intensive Care, Cambridge